CLINICAL TRIAL: NCT02066493
Title: Giant Intracranial Aneurysm Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. med. Julius Dengler (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Julius Dengler, MD, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: Giant; CS-2009-13 (Other Grant/Funding Number: Center for Stroke Research - Berlin)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Intracranial Aneurysms
Keywords: giant intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- conservative management: neither surgical nor endovascular management
- endovascular management: endovascular management
- surgical management: surgical management

SUMMARY:
The purpose of this study is to generate detailed insight into which therapies of giant intracranial aneurysms are being conducted, to document the natural history and the outcome of treatment over 5 years after inclusion into the Registry and to follow imaging data of giant aneurysms over years after diagnosis.

DETAILED DESCRIPTION:
Definition of aims, eligibility of patients and data flow

In August 2009 a steering committee was appointed and its first meeting took place in Berlin. Here the aims of the registry were defined as follows: 1) To generate detailed insight into which therapies are being conducted. 2) To document the natural history of patients and follow it over years after diagnosis. 3) To follow imaging data of giant aneurysms over years after diagnosis, whether treated conservatively or not. 4) To expand the register into several disciplines (by inviting neuroradiologic and neurologic centers to join) and internationally.

Inclusion criteria are a) the diagnosis of a giant intracranial aneurysm by CT, MRI or regular angiography, b) age 18 years and older and c) informed consent. There are no exclusion criteria. If a patient is not able to give informed consent due to his or her clinical situation, the legal representative of the patient (e.g. family member) will be informed and asked to sign the consent form on behalf of the patient.

Patients are recruited consecutively in responsibility of each center. In addition to the prospective part there is a retrospective part in which patients are included that were admitted after January 2006. Data are gathered at admission, discharge and 1/3/5 years after discharge. Starting from February 2010 a 9-month pilot phase was conducted in order to identify and correct possible problems of data acquisition.

Development of a study protocol

Relevant variables were discussed on the basis of existing literature on giant intracranial aneurysms. All variables were chosen so that they can be determined in a routine clinical context even in small centers with minimal technical equipment. Data collection was decided to be carried out using a modular structure, consisting of a basic module and additional modules for specific research questions.

The steering committee decided on the content of a mandatory basic data collection for all centers. This basic module was designed to keep the amount of variables at a minimum so that data collection can be conducted as safely and quickly as possible by physicians of all disciplines. It focuses on the clinical course between initial presentation and discharge but also includes data on patient history, such as risk factors and possible prior aneurysm therapy. A neurological examination of cranial nerve functions, motor capability and speech is conducted initially, at discharge and during 3 mandatory follow-up examinations. At each examination the patients' physical condition is recorded using internationally accepted and reliable grading systems. The investigator is asked to not only record a clinical diagnosis, such as epileptic seizure or incidental finding, but also use imaging data to produce a radiological diagnosis and characterize the aneurysm regarding its location, size, shape and structure. The mode of therapy is documented choosing between conservative, surgical and endovascular options and combinations thereof. Possible complications are recorded as well as radiologic results of intervention.

Each center is given the option to take part in additional extra modules, which serve as a basis for spin-off projects resulting from the discussion within the study group. This comprises for example an imaging module to lead to a better understanding of how giant intracranial aneurysms develop over time. It will monitor changes in aneurysm configuration and flow dynamics using 3D-imaging data. A cost module will integrate data on treatment expenses making it possible to compare the costs of each mode of therapy.

An external review of the study protocol was conducted to ensure high methodological quality and wide acceptance of the results. For this purpose a preliminary working report was forwarded to 4 independent experts in the field of neurovascular research. The reviewers were asked to comment on the appropriateness of the methods, the practicability of our variables and the coverage of relevant aspects of giant intracranial aneurysm care. The comments of the external reviewers were gathered and discussed within the steering committee. Based on the recommendations of the external reviewers, a final revision of the study protocol took place.

Primary hypothesis, study outcome and statistical analyses

The primary hypothesis of the study is that conservative, endovascular and surgical therapy result in equal aneurysm rupture rates. Therefore primary outcome will be aneurysm rupture rate at 5 years of follow up.

The sample size calculation is based on the estimated 5-year cumulative rupture rates for patients with unruptured giant aneurysm given in the ISUIA-Trial. According to their results we assume a 5-year rupture rate of 0.30 irrespective of which specific treatment is applied. Because of a lack of data on special rupture rates regarding patients treated with the three considered methods, sample size calculation was done for one proportion based on precision analysis. Consequently, a two-sided 95% confidence interval with a width equal to 0.10 is achieved by a sample size of 320 patients. For the outcomes death or rupture the corresponding survival functions with 95% confidence intervals will be estimated by the Kaplan-Meier method. The null-hypotheses of equal survival curves for two treatment groups will be tested by the Log-Rank test. With documented dates of rupture events the sample size of 320 calculated above is sufficient to detect moderate effects of possible predictors for rupture by Cox proportional hazards regression within a secondary analysis. Furthermore we can model the logit of rupture after 5 years by binary logistic regression detecting possible moderate to considerable effects of predictors. Therapy (conventional, surgery or endovascular) will be the main factor of interest for both multivariable analyses.

Patient recruitment / Data storage / Quality assurance

In 2008 patient recruitment began at the Charité Berlin, one year later data from other centers were included as well, initially only in Germany, later on throughout Europe and Japan. Patient data are stored using pseudonyms. Centers can either use a fax-based data inclusion form or a web-based entry form. All data are stored at the Charité - Berlin. For quality assurance a monitoring visit to the 7 most-including centers was conducted in 2013.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of a giant intracranial aneurysm

Exclusion Criteria:

* age younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2008-12-05 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
aneurysm rupture rate - diagnosed radiologically (e.g. by CT) or clinically | 5 years

SECONDARY OUTCOMES:
health status of the patient quantified by modified Rankin Scale in combination with a basic neurological exam | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Julius Dengler, MD, Study Chair — Charite University, Berlin, Germany; Peter Vajkoczy, Prof., MD, Study Director — Charite University, Berlin, Germany; Veit Rohde, Prof., MD, Study Director — University of Goettingen; Peter Heuschmann, Prof., MD, Study Director — University of Wuerzburg; Bernhard Meyer, Prof., MD, Study Director — Technical University of Munich; Daniel Ruefenacht, Prof., MD, Study Director — Klinikum Hirslanden Zurich; Matthias Endres, Prof., MD, Study Director — Charite University, Berlin, Germany
Locations (23):
- Department of Neurosurgery, Medical University Vienna, Vienna, Austria
- Department of Neurosurgery, Helsinki University Central, Helsinki, Finland
- Department of Neuroradiology, University Hospital, Toulouse, France
- Germany (12):
  - Department of Neurology - Charité Berlin, Berlin
  - Department of Neurosurgery, Charité Berlin, Berlin
  - Department of Neurosurgery and Neuroradiology, Klinikum Deggendorf, Deggendorf
  - Department of Neurosurgery, University of Freiburg, Freiburg im Breisgau
  - Department of Neurosurgery - University of Goettingen, Göttingen
  - Department of Neurosurgery - University of Greifswald, Greifswald
  - Department of Neurosurgery - University of Hamburg, Hamburg
  - Department of Neurosurgery, Friedrich-Schiller-University, Jena
  - Department of Neuroradiology, University of Leipzig, Leipzig
  - Department of Neurosurgery - Technical University of Munich, Munich
  - Department of Neurosurgery - University of Regensburg, Regensburg
  - Institut für Klinische Epidemiologie und Biometrie der Universität Wuerzburg, Würzburg
- Department of Neuroradiology, Ospedale Niguarda Ca' Granda, Milan, Italy
- Department of Neurosurgery, Jikei University, Tokyo, Japan
- Department of Neurosurgery, University Hospital, Utrecht, Netherlands
- Department of Neurosurgery, Burdenko Neurosurgical Institute, Moscow, Russia
- Switzerland (4):
  - Department of Neurosurgery, Kantonsspital Aarau, Aarau
  - Department of Neurosurgery - University of Geneva, Geneva
  - Department of Neuroradiology - Klinikum Hirslanden, Zurich
  - Department of Neurosurgery, University Hospital of Zurich, Zurich

REFERENCES:
- [Background] Dengler J, Heuschmann PU, Endres M, Meyer B, Rohde V, Rufenacht DA, Vajkoczy P; Giant Intracranial Aneurysm Study Group. The rationale and design of the Giant Intracranial Aneurysm Registry: a retrospective and prospective study. Int J Stroke. 2011 Jun;6(3):266-70. doi: 10.1111/j.1747-4949.2011.00588.x. Epub 2011 Apr 7. PMID 21557815
- [Derived] Dengler J, Rufenacht D, Meyer B, Rohde V, Endres M, Lenga P, Uttinger K, Rucker V, Wostrack M, Kursumovic A, Hong B, Mielke D, Schmidt NO, Burkhardt JK, Bijlenga P, Boccardi E, Cognard C, Heuschmann PU, Vajkoczy P. Giant intracranial aneurysms: natural history and 1-year case fatality after endovascular or surgical treatment. J Neurosurg. 2019 Dec 6;134(1):49-57. doi: 10.3171/2019.8.JNS183078. Print 2021 Jan 1. PMID 31812141
- [Derived] Haemmerli J, Lenga P, Hong B, Kursumovic A, Maldaner N, Burkhardt JK, Bijlenga P, Rufenacht DA, Schmidt NO, Vajkoczy P, Dengler J. Clinical implications and radiographic characteristics of the relation between giant intracranial aneurysms of the posterior circulation and the brainstem. Acta Neurochir (Wien). 2019 Sep;161(9):1747-1753. doi: 10.1007/s00701-019-04016-x. Epub 2019 Jul 29. PMID 31359190
- [Derived] Lenga P, Hohaus C, Hong B, Kursumovic A, Maldaner N, Burkhardt JK, Bijlenga P, Rufenacht DA, Schmidt NO, Vajkoczy P, Dengler J. Giant intracranial aneurysms of the posterior circulation and their relation to the brainstem: analysis of risk factors for neurological deficits. J Neurosurg. 2019 Aug 1;131(2):403-409. doi: 10.3171/2018.4.JNS172343. Epub 2018 Aug 10. PMID 30095339
- [Derived] Durner G, Piano M, Lenga P, Mielke D, Hohaus C, Guhl S, Maldaner N, Burkhardt JK, Pedro MT, Lehmberg J, Rufenacht D, Bijlenga P, Etminan N, Krauss JK, Boccardi E, Hanggi D, Vajkoczy P, Dengler J; Giant Intracranial Aneurysm Study Group. Cranial nerve deficits in giant cavernous carotid aneurysms and their relation to aneurysm morphology and location. Acta Neurochir (Wien). 2018 Aug;160(8):1653-1660. doi: 10.1007/s00701-018-3580-2. Epub 2018 Jun 9. PMID 29948299
- [Derived] Maldaner N, Guhl S, Mielke D, Musahl C, Schmidt NO, Wostrack M, Rufenacht DA, Vajkoczy P, Dengler J; Giant Intracranial Aneurysm Study Group. Changes in volume of giant intracranial aneurysms treated by surgical strategies other than direct clipping. Acta Neurochir (Wien). 2015 Jul;157(7):1117-23; discussion 1123. doi: 10.1007/s00701-015-2448-y. Epub 2015 May 23. PMID 26002711
- [Derived] Dengler J, Maldaner N, Bijlenga P, Burkhardt JK, Graewe A, Guhl S, Hong B, Hohaus C, Kursumovic A, Mielke D, Schebesch KM, Wostrack M, Rufenacht D, Vajkoczy P, Schmidt NO; Giant Intracranial Aneurysm Study Group. Perianeurysmal edema in giant intracranial aneurysms in relation to aneurysm location, size, and partial thrombosis. J Neurosurg. 2015 Aug;123(2):446-52. doi: 10.3171/2014.10.JNS141560. Epub 2015 Apr 17. PMID 25884259
- [Derived] Dengler J, Maldaner N, Bijlenga P, Burkhardt JK, Graewe A, Guhl S, Nakamura M, Hohaus C, Kursumovic A, Schmidt NO, Schebesch KM, Wostrack M, Vajkoczy P, Mielke D; Giant Intracranial Aneurysm Study Group. Quantifying unruptured giant intracranial aneurysms by measuring diameter and volume--a comparative analysis of 69 cases. Acta Neurochir (Wien). 2015 Mar;157(3):361-8; discussion 368. doi: 10.1007/s00701-014-2292-5. Epub 2014 Dec 12. PMID 25502806
- See also: CSB - Center for Stroke Research - Berlin — http://www.schlaganfallcentrum.de